CLINICAL TRIAL: NCT05363007
Title: Spleen Irradiation With Nanoliposomal Irinotecan Plus 5-FU and Leucovorin in Metastatic Pancreatic Adenocarcinoma: a Phase II Study (SINAI)
Brief Title: Spleen Irradiation With Nanoliposomal Irinotecan Plus 5-FU and Leucovorin in Metastatic Pancreatic Adenocarcinoma
Acronym: SINAI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202110064MIPB
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-06

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: pancreatic cancer; nanoliposomal irinotecan; spleen irradiation
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — irinotecan sucrosofate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Upfront SI (Experimental): Upfront nanoliposomal irinotecan + 5-FU/leucovorin plus SI
  Interventions: Drug: nanoliposomal irinotecan; Radiation: spleen irradiation
- Add-on SI (Experimental): Add-on SI following limited progression to nanoliposomal irinotecan + 5-FU/leucovorin
  Interventions: Drug: nanoliposomal irinotecan; Radiation: spleen irradiation

INTERVENTIONS:
Drug: nanoliposomal irinotecan — Upfront SI (Arm A): Upfront nanoliposomal irinotecan (80 mg/m2, day 1) + 5-FU/leucovorin (2400 mg/m2, 400 mg/m2) plus SI
  Add-on SI (Arm B): Add-on SI following limited progression to prior nanoliposomal irinotecan (last dose used) + 5-FU/leucovorin (last dose used)
  Other Names: 5-FU/leucovorin
Radiation: spleen irradiation — Upfront SI (Arm A): upfront spleen irradiation (1 Gy/fx, day 1-4) in cycle 2
  Add-on SI (Arm B): add-on spleen irradiation (1 Gy/fx, day 1-4) in cycle 1 following limited progression to prior nanoliposomal irinotecan + 5-FU/leucovorin

SUMMARY:
Splenomegaly is common in advanced pancreatic ductal adenocarcinoma (PDAC). The spleen is an important source of immune suppressive cells and phagocytic cells and may mediate the accumulation of liposomal drugs and immunosuppression. In this study, spleen irradiation (SI) will be added to standard chemotherapy.

DETAILED DESCRIPTION:
Splenomegaly is common in PDAC. Therefore, we design a phase II study to enroll metastatic PDAC patients who have failed prior gemcitabine-based therapy and have splenomegaly. With add-on SI to standard nal-IRI/FL therapy, we hypothesize that 1) splenic phagocytes and spleen volume will be reduced with attenuated entrapment of nal-IRI within spleen, 2) splenic source of immunosuppressive immune cells will be reduced with potential reconstitution of antitumor TME.

ELIGIBILITY:
Inclusion Criteria:

* Arm A:
* histologically or cytologically proved PDAC
* metastatic PDAC
* failed frontline gemcitabine-based chemotherapy and preparing for application of NHI-reimbursed nal-IRI/FL
* splenomegaly: SV > 270 ml (estimated)
* lymphopenia: < 1200/mm3
* no previous radiotherapy, local therapy (eg. radiofrequency ablation, irreversible electroporation, etc.), cell therapy (autologous or allogenic) used for pancreatic cancer
* presence of at least one measurable lesion outside spleen
* age between 20 and 75 years at registration
* ECOG performance status of 0 or 1
* adequate major organ functions
* Arm B:
* limited progressive disease after prior nal-IRI/FL
* prior treatment of nal-IRI/FL at least 4 doses
* histologically or cytologically proven PDAC
* metastatic PDAC before starting prior nal-IRI/FL
* failed frontline gemcitabine-based chemotherapy before prior nal-IRI/FL
* presence of at least one measurable lesion outside spleen
* age between 20 and 75 years at registration
* ECOG performance status of 0 or 1 or 2 after the chemotherapy phase
* adequate major organ functions

Exclusion Criteria:

* interstitial lung disease
* presence of diarrhea ≥ CTCAE v.5.0 grade 2
* concomitant systemic infection requiring treatment
* clinically significant co-morbid medical conditions
* prior organ allograft or allogeneic bone marrow transplantation
* received systemic corticosteroids or immunosuppressants within 28 days before registration
* known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome
* moderate or severe ascites, pleural effusion, or pericardial effusion requiring treatment
* central nervous system metastasis
* prior or concurrent malignancies within the last 3 years, with the exception of carcinoma in situ of the cervix, or basal type skin cancer
* any major surgery within 4 weeks of study treatment. Participants must have recovered from the effects of major surgery or significant traumatic injury.
* pregnant women or nursing mothers, or positive pregnancy tests
* severe mental disorder
* spleen metastasis or direct invasion

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
12W-PFS | 12 week
  12-week PFS rate (%)

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Hung Yang, MD., PhD., Principal Investigator — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No